CLINICAL TRIAL: NCT02241551
Title: Phase II Study of Neoadjuvant Chemotheraphy (Gemcitabine and Nab-Paclitaxel vs. mFOLFIRINOX) and Sterotatic Body Radiation Therapy for Borderline Resectable Pancreatic Cancer
Brief Title: Phase II Neoadjuvant Chemotheraphy (Gemcitabine and Nab-Paclitaxel vs. mFOLFIRINOX) and Sterotatic Body Radiation Therapy for Borderline Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated with the IRB ended early as logistical concerns of the SBRT
Sponsor: Nathan Bahary, MD (Other)
Responsible Party: Sponsor-Investigator, Nathan Bahary, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 13-143
Record Dates: First submitted 2014-08-29; First posted 2014-09-16 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Borderline Resectable Pancreatic Cancer
Keywords: Borderline; Resectable; Pancreatic; Cancer; Neoadjuvant; Chemotheraphy; Gemcitabine; Nab-Paclitaxel; mFOFIRINOX; Sterotatic Body Radiation Therapy
MeSH Terms: conditions — Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel; Irinotecan; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemcitabine/nab-paclitaxel (Experimental): three cycles of treatment in the gemcitabine/nab-paclitaxel
  Interventions: Drug: gemcitabine/nab-paclitaxel
- mFOLFIRINOX (Experimental): 6 cycles in the mFOLFIRINOX
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: gemcitabine/nab-paclitaxel — three cycles of treatment in the gemcitabine/nab-paclitaxel
  Other Names: Gemzar; ABRAXANE
  Arms: gemcitabine/nab-paclitaxel
Drug: mFOLFIRINOX — 6 cycles in the mFOLFIRINOX
  Other Names: irinotecan; fluorouracil; oxaliplatin
  Arms: mFOLFIRINOX

SUMMARY:
This is a prospective, randomized phase II trial. Patients diagnosed with borderline resectable pancreatic adenocarcinoma will be randomly assigned to one of two treatment arms, either mFOLFIRINOX or gemcitabine and nab-paclitaxel. After three cycles of treatment in the gemcitabine/nab-paclitaxel arm and 6 cycles in the mFOLFIRINOX arm, patients will be restaged with CT scans and if they remain borderline resectable or have improvement of their disease They will then proceed to SBRT followed by surgical resection.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following criteria within 28 days of randomization (unless otherwise indicated) to be enrolled in the protocol:

* Histologically or cytologically proven adenocarcinoma of the pancreas. If the patient has mixed tumor with predominant adenocarcinoma pathology, they can be enrolled.
* Subjects will be staged according to the 2010 American Joint Committee on Cancer (AJCC) staging system with pathologic stage T1-4, N0 being eligible; and have a primary tumor of the pancreas (either pancreatic head, neck, uncinate process, or body/tail)
* The tumor must be deemed as being borderline resectable. Final CT confirmation of surgical staging/ eligibility will be at the discretion of the pancreatic surgeon of the patient.
* Disease is confined to locoregional site as confirmed by the CT and / or diagnostic staging laparoscopy to avoid occult peritoneal deposits. Diagnostic laproscopy will be only if absolutely required
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) on imaging studies CT
* Screening Endoscopic ultrasound if done prior to consent but within 6 weeks of expected randomization date it may be used.
* Karnofsky performance status greater than or equal to 70 or Eastern Cooperative Oncology Group (ECOG) performance of 0-2.
* Age > 18
* Estimated life expectance > 12 weeks
* If female patient is of child bearing potential, she must have a negative serum pregnancy test (βhCG) documented up to 72hrs prior to administration of first study drug
* Patient has screening blood work performed which includes the following (should be drawn ≤ 14 days prior to randomization)
* absolute neutrophil count (ANC) > 1.5 x 109/L
* Platelet count ≥ 100000/mm3
* Hemoglobin (HgB) ≥ 9g/dL
* aspartate aminotransferase (AST),Alanine Aminotransferase (ALT)≤ 2.5 x upper limit of normal (ULN) Total Bilirubin ≤ ULN
* Serum Cr within normal limits (WNL)
* Coagulation studies with Prothrombin Time and International Normalized Ratio (PT/INR) and partial thromboplastin time (PTT) within normal limits (±15%). • Patient has a urinalysis obtained (≤14 days prior to randomization) and the results are deemed not clinically significant by the investigator.
* Patient has no evidence of jaundice at the time of enrolment. If stent is required to alleviate jaundice, it should be metallic. If patient has a previously placed stent and this is plastic, this should be changed to metallic.
* Patient's pain symptoms have remained stable with no adjustment to analgesics within 7 days prior to randomization. Patient must be able to swallow entreat medications with no requirement for a feeding tube. Patient's must not have intractable nausea or vomiting which prohibits the patient from oral medications
* Diabetes must be controlled prior to enrollment
* Disease must be encompassed in a reasonable SBRT "portal" as defined by the treating radiation oncologist

Exclusion Criteria:

* Ineligible Histology including non-adenocarcinomas, adenosquamous carcinoma, islet cell carcinomas, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct and ampullary carcinomas
* Evidence of distant metastasis on upright chest x-ray, CT or other staging studies
* Subjects with recurrent disease
* Prior radiation therapy to the upper abdomen or liver at the discretion of the treating radiation oncologist could impair delivery of the prescribed radiation treatment
* Prior chemotherapy
* Subjects in their reproductive age who are breast feeding or have a positive pregnancy test
* Any co-morbid condition of sufficient severity to limit full compliance with the protocol per assessment by the individual treating physician
* Concurrent active infection
* Previous or current malignancies of other histologies within the last 3 yrs prior to randomization; with the exception of cervical cancer in situ, adequately treated basal cell or squamous cell carcinoma of skin or treated low risk prostate cancer
* Patient with known historical or active infection with HIV, Hepatitis B or Hepatitis C
* Patient who has undergone recent major surgery, other than diagnostic surgical procedure within 4 weeks prior to randomization.
* Patient who has a history of allergy or hypersensitivity to any of the study drugs.
* Patients with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, interstitial pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies
* Patients with greater than 2 screening peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine/Nab-paclitaxel: Patients that received three cycles of treatment in the gemcitabine/nab-paclitaxel
- mFOLFIRINOX: Patients that received 6 cycles in the mFOLFIRINOX
Period: Overall Study
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants analyzed or is zero for the Treatment Arm in which zero participants were treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 54 [54 to 54] |  | 54 [54 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy Using Neo-adjuvant Gemcitabine Plus Nab-paclitaxel in Patients Receiving SBRT and Surgery for Borderline Resectable Pancreatic Cancer, Using Neo-adjuvant mFOLFIRINOX as a Control
Description: Efficacy: pathological complete response (pCR) and R0 resection. Safety: Grade 4 toxicity.
Time Frame: up to 5 years
Population: Patient did not receive three cycles of treatment - data were not collected.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: R0 Resection Rates in Borderline Resectable Pancreatic Cancer
Time Frame: Up to 5 years
Population: Patient did not receive three cycles of treatment - data were not collected.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Grade 3 and 4 Toxicities for the 2 Chemotherapy Regimens That Occur After Cycle 1 Day 1
Description: According to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTAE, v4.0)
Time Frame: Up to 5 years
Population: Patient was not treated - no data collected.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Ca19-9 Response to Neoadjuvant Chemotherapy
Time Frame: Up to 5 years
Population: Patient did not receive three cycles of treatment - data were not collected / zero total participants were analyzed.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Disease Progression
Time Frame: Up to 5 years
Population: Patient did not receive three cycles of treatment - data not collected.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Measurement of Biomarkers (SPARC, RM1 and SMAD4) in Tissues
Description: This wil be measured in tissues that are obtained at screening and in the resected tumour specimen
Time Frame: Up to 5 years
Population: Patient did not receive three cycles of treatment - data not collected.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Radiological Response Rate to Therapy
Description: Radiological improvements will be evaluated by determining changes in density of measurable disease on CT scan pre and post chemotherapy
Time Frame: Up to 5 years
Population: Patient did not receive three cycles of treatment - data not collected.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Quality of Life Effects of Chemotherapy on Patients Receiving Chemotherapy and SBRT
Description: This will be measured using the FACT-HB questionaire
Time Frame: Up to 5 years
Population: Patient did not receive three cycles of treatment - data not collected.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The number of participants at risk for Serious Adverse Events is zero for the Treatment Arm in which zero participants were treated.
  The number of participants at risk for Other (Not Including Serious) Adverse Events is zero for the Treatment Arm in which zero participants were treated.
  The number of participants at risk for All-Cause Mortality is zero for the Treatment Arm in which zero participants were treated.
Arm/Group | Gemcitabine/Nab-paclitaxel | mFOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Nab-paclitaxel (N=1) | mFOLFIRINOX (N=0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT02241551/Prot_SAP_000.pdf